CLINICAL TRIAL: NCT00310752
Title: Evaluation of DermStream(tm) - an Irrigation Product for Chronic Wound Management
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EnzySurge (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS-1
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Venous Insufficiency; Diabetes
MeSH Terms: conditions — Venous Insufficiency; Diabetes Mellitus

INTERVENTIONS:
Device: DermaStream(tm) application and Streaming of Saline

SUMMARY:
The primary purpose of this study is to evaluate the safety of DermaStream(tm) in the management of chronic wounds.

Other goals of this study are to gain feedback from patients and healthcare providers on the ease of use (the ergonomic aspect) of the device, and to make a preliminary evaluation of the efficacy of DermaStream(tm) in chronic wound management.

DETAILED DESCRIPTION:
Until now no expected or unexpected adverse events were occurred

ELIGIBILITY:
Inclusion Criteria:

* Diabetic ulcer, OR Venous insufficiency ulcer
* Age range: 18-80 years
* Wound max. diameter range: 1.5 - 10 centimeters
* Wound San Antonio assessment system: grade 1 and 2, stage A and B
* Palpable pulses in the Posterior Tibial and the Dorsalis Pedis arteries
* Ankle-Brachial Index > 0.7 by Doppler
* Wound present for at least 6 weeks
* Wound location: foot or calf, at a location where the device can be attached properly
* Lack of purulent discharge from the wound.

Exclusion Criteria:

* Hypoalbuminemia: Albumin < 2gr/dl
* Right-side congestive heart failure with edema of legs: +2 or higher
* Renal insufficiency: Cr > 2 mg/dl
* Abnormal liver function: ALT or AST>300
* Skin disorders adjacent to the wound, unrelated to the pathology of the wound
* Non-cooperative patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arie Bass, Prof., Principal Investigator — Asaf Harofe Medical Center
Locations (1):
- Vascular Surgery Department, Asaf Harofe Medical Center, Zrifin, Israel